CLINICAL TRIAL: NCT04400877
Title: Prevalence and Severity of Venous Thromboembolism in a General Population During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, MD, Emergency department head of research, University Hospital, Linkoeping
Other Study IDs: SE2020-02701
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Venous Thromboembolism; Pulmonary Embolism; Deep Vein Thrombosis; SARS-CoV 2
MeSH Terms: conditions — COVID-19; Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 pos: Patients who have been tested positive for SARS-CoV-2 virus by either nasopharyngeal swab PCR or antibody testing.
  Interventions: Diagnostic Test: Diagnostic examination for venous thromboembolism
- SARS-CoV-2 neg: Patients without symptoms for SARS-CoV-2 infection who haven't been tested for the virus or patients with symptoms who have been tested negative for SARS-CoV-2 virus by either nasopharyngeal swab PCR or antibody testing.
  Interventions: Diagnostic Test: Diagnostic examination for venous thromboembolism

INTERVENTIONS:
Diagnostic Test: Diagnostic examination for venous thromboembolism — Patients who have done a diagnostic examination for suspected VTE (pulmonary embolism och deep venous thrombosis) within the health care system of Region Östergötland. Patients without matching diagnostic examination but with a new diagnosis of pulmonary embolism or deep venous thrombosis during the same time periods will also be taking into account.
  Other Names: CT Pulmonary Angiogram (CTPA); Ultrasound for deep venous thrombosis (DVT)

SUMMARY:
The purpose of this study is to investigate the prevalence of venous thromboembolism in a regional health care system (Region Östergötland, Sweden) before and during the SARS-COV-2 pandemic. In a retrospective observational study, we will review patient data, diagnostic data and treatment data over a three-month period since the onset of the SARS-COV-2 pandemic. This data will be compared with data from the corresponding time frame during the years 2015 to 2019.

DETAILED DESCRIPTION:
In the current SARS-COV-2 pandemic there is a concern about an increased risk of venous thromboembolism (VTE) concurrent with the infection, including both pulmonary embolism (PE) and deep venous thrombosis (DVT) (Klok et al. 2020; Cui et al. 2020; Helms et al. 2020; Leonard-Lorant et al. 2020; Poissy et al. 2020). International guidelines now recommend prophylactic anticoagulation for all hospitalized patients with a SARS-COV-2 infection in the absence of any contraindication (Thachil et al. 2020). The majority of the studies on VTE in SARS-COV-2 infections have been carried out in the ICU and show prevalence of VTE of between 20 and 30%.(Klok et al. 2020; Cui et al. 2020; Helms et al. 2020). This is a clear increase compared to the less than 10 % prevalence seen in other ICU patients (Muscedere, Heyland, and Cook 2007; Deborah Cook et al. 2005; D. Cook et al. 2000). However, a single center study on consecutive ICU patients with severe sepsis showed a prevalence of VTE of 37% (Kaplan et al. 2015) and another recent publication of patients with severe influenza A/H1N1 infection had a prevalence of VTE of 44% (Obi et al. 2019).

This raises the question whether the increase in VTE seen in recent publications of SARS-COV-2 infections is the result of the specific pathophysiology of the virus itself or the subsequent sepsis with multiorgan failure seen in most complicated and severe cases. The former would have large implications for patients treated outside the ICU and possibly outside hospitals (Thachil et al. 2020).

The aim of this study will be to investigate the prevalence of VTE in a regional healthcare system prior to, and during the SARS-COV-2 pandemic and the differences between ICU, hospitalized and outpatient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that has done a Computer Tomography Angiography of the lungs between 1:st of March and 31:st of May each year from 2015 to 2020
* Any patient that has done a Ultrasound of the legs between 1:st of March and 31:st of May each year from 2015 to 2020
* Any patient with a new diagnosis of pulmonary embolism or deep venous thrombosis between 1:st of March and 31:st of May each year from 2015 to 2020

Exclusion Criteria:

* Incomplete diagnostic examination
* Follow-up examination of know acute VTE
* Primary investigation done outside the healthcare system
* Patient <18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For enrolment, we will consider all patients who have done a diagnostic examination for suspected VTE (pulmonary embolism och deep venous thrombosis) within the health care system of Region Östergötland during March, April and May 2015 through 2020. We will also include all patients with a new diagnosis of pulmonary embolism or deep venous thrombosis during the same time periods.
  Region Östergötland/Östergötland County has a population of 465,495 (December 31, 2019).
Sampling Method: Probability Sample
Enrollment: 7795 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Is there an increased prevalence of venous thromboembolism in a regional healthcare system in Sweden during the SARS-CoV-2 pandemic? | March to May in 2020
Is a SARS-CoV-2-infection an isolated risk factor for thromboembolism? | March to May in 2020

SECONDARY OUTCOMES:
Are there geographic differences in the prevalence of venous thromboembolism within the healthcare system? | March to May in 2020
Is venous thromboembolism associated with increased mortality adjusted for relevant comorbidities? | March to May in 2020
How long is the time between symptom onset of the SARS-CoV-2-infection and any subsequent venous thromboembolism? | March to May in 2020
Is treatment with prophylactic antithrombotic or anticoagulant treatment associated with increased survival? | March to May in 2020

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wretborn, MD, Principal Investigator — Emergency Department, University Hospital Linköping, Sweden; Patrik Benjaminsson Nyberg, PhD, Principal Investigator — Emergency Department, University Hospital Linköping, Sweden; Matthias Jörg, MD, Principal Investigator — Emergency Department, University Hospital Linköping, Sweden
Locations (1):
- University Hospital Linköping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cook D, Attia J, Weaver B, McDonald E, Meade M, Crowther M. Venous thromboembolic disease: an observational study in medical-surgical intensive care unit patients. J Crit Care. 2000 Dec;15(4):127-32. doi: 10.1053/jcrc.2000.19224. PMID 11138871
- [Background] Cook D, Crowther M, Meade M, Rabbat C, Griffith L, Schiff D, Geerts W, Guyatt G. Deep venous thrombosis in medical-surgical critically ill patients: prevalence, incidence, and risk factors. Crit Care Med. 2005 Jul;33(7):1565-71. doi: 10.1097/01.ccm.0000171207.95319.b2. PMID 16003063
- [Background] Cui S, Chen S, Li X, Liu S, Wang F. Prevalence of venous thromboembolism in patients with severe novel coronavirus pneumonia. J Thromb Haemost. 2020 Jun;18(6):1421-1424. doi: 10.1111/jth.14830. Epub 2020 May 6. PMID 32271988
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Background] Kaplan D, Casper TC, Elliott CG, Men S, Pendleton RC, Kraiss LW, Weyrich AS, Grissom CK, Zimmerman GA, Rondina MT. VTE Incidence and Risk Factors in Patients With Severe Sepsis and Septic Shock. Chest. 2015 Nov;148(5):1224-1230. doi: 10.1378/chest.15-0287. PMID 26111103
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Leonard-Lorant I, Delabranche X, Severac F, Helms J, Pauzet C, Collange O, Schneider F, Labani A, Bilbault P, Moliere S, Leyendecker P, Roy C, Ohana M. Acute Pulmonary Embolism in Patients with COVID-19 at CT Angiography and Relationship to d-Dimer Levels. Radiology. 2020 Sep;296(3):E189-E191. doi: 10.1148/radiol.2020201561. Epub 2020 Apr 23. PMID 32324102
- [Background] Muscedere JG, Heyland DK, Cook D. Venous thromboembolism in critical illness in a community intensive care unit. J Crit Care. 2007 Dec;22(4):285-9. doi: 10.1016/j.jcrc.2007.02.003. Epub 2007 Jul 5. PMID 18086398
- [Background] Poissy J, Goutay J, Caplan M, Parmentier E, Duburcq T, Lassalle F, Jeanpierre E, Rauch A, Labreuche J, Susen S; Lille ICU Haemostasis COVID-19 Group. Pulmonary Embolism in Patients With COVID-19: Awareness of an Increased Prevalence. Circulation. 2020 Jul 14;142(2):184-186. doi: 10.1161/CIRCULATIONAHA.120.047430. Epub 2020 Apr 24. No abstract available. PMID 32330083
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Derived] Wretborn J, Jorg M, Benjaminsson Nyberg P, Wilhelms DB. Risk of venous thromboembolism in patients with COVID-19 during 2020; a retrospective cross-sectional study in a Swedish health care system. Sci Rep. 2023 Apr 4;13(1):5469. doi: 10.1038/s41598-023-32637-x. PMID 37015984
- See also: Complete study protocol as used for approval at the Swedish Ethical Review Authority — https://docs.google.com/document/d/1rNUhsHak2dVSHrG0Hz6bV7TVgcdyNc6hGXjrhCOx7HU/edit?usp=sharing